CLINICAL TRIAL: NCT01987999
Title: Phase II Eradication of Prostate Cancer Using F-989
Brief Title: Eradication of Prostate Cancer Using F-989
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Optimal Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-9892131
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Acetogenins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acetogenins (Experimental): Acetogenins twice (BID) per day for 12 months
  Interventions: Dietary Supplement: Acetogenins

INTERVENTIONS:
Dietary Supplement: Acetogenins

SUMMARY:
The purpose of this study is to confirm the findings of an early study with prostate cancer and to expand our knowledge of treating prostate cancer using F-989.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of prostate cancer
* Referred to the study by their treating physician

Exclusion Criteria:

- Any type of treatment before starting study

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Gleason Score | 1 year
  A Gleason Score is obtained from the results of a transrectal needle biopsy of the prostate.

SECONDARY OUTCOMES:
Prostate Specific Antigens (PSA) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steven Osguthorpe, ND, Principal Investigator — Optimal Health Research